CLINICAL TRIAL: NCT06244251
Title: Comparison of Operational Outcomes and Long-term Benefits Between Laparoendoscopic Single-site Surgery and Multi-port Laparoscopy in Treating Uterine Fibroids
Brief Title: Comparison Between Laparoendoscopic Single-site Surgery and Multi-port Laparoscopy in Treating Uterine Fibroids
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West China Second University Hospital (Other)
Responsible Party: Principal Investigator, Zheng Ying, Dean, Department of Obstetrics and Gynecology, West China Second University Hospital, Sichuan University, West China Second University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023YFS0046
Record Dates: First submitted 2023-08-09; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: Uterine Fibroid; Uterine Sarcoma; Uterine Leiomyosarcoma
Keywords: Uterine fibroids; TU-LESS; Multi-port laparoscopic surgery
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TU-LESS for myomectomy (Experimental): Patients complaint of symptoms resulting from uterine fibroids, such as abnormal vaginal bleeding, frequent micturition, lower abdominal pain, constipation, etc or patients with uterine fibroids which were identified accidentally during routine body examination who consulted at our center for surgical removal of the fibroids. In the meantime, the diagnosis of uterine fibroids should be reconfirmed by at least one radiological examination at our center. The patients in the experiment group were those who received transumbilical laparoendoscopic single site surgery (TU-LESS) for myomectomy.
  Interventions: Procedure: TU-LESS
- MPLS for myomectomy (Active Comparator): Patients complaint of symptoms resulting from uterine fibroids, such as abnormal vaginal bleeding, frequent micturition, lower abdominal pain, constipation, etc or patients with uterine fibroids which were identified accidentally during routine body examination who consulted at our center for surgical removal of the fibroids. In the meantime, the diagnosis of uterine fibroids should be reconfirmed by at least one radiological examination at our center. The patients in the experiment group were those who received multiport laparoscopic surgery (MPLS) for myomectomy.
  Interventions: Procedure: MPLS

INTERVENTIONS:
Procedure: TU-LESS — TU-LESS group will receive TU-LESS for myomectomy; MPLS group will receive MPLS for myomectomy
  Arms: TU-LESS for myomectomy
Procedure: MPLS — Patients with uterine who plan to receive MPLS for myomectomy
  Arms: MPLS for myomectomy

SUMMARY:
Myomectomy was preferably applied in females with reproductive requirements, which could be achieved by transumbilical laparoendoscopic single-site surgery (TU-LESS) or multi-port laparoscopic surgery (MPLS). Power morcellation used in MPLS was correlated with unidentified risk of tumor dissemination, especially in cases with accidental surgical findings of uterine sarcoma or leiomyosarcoma. Moreover, TU-LESS was reported to exceed MPLS in fast recovery. Therefore, the aim of this prospective cohort study is to compare the effectiveness of fast recovery and relative risk of tumor dissemination between TU-LESS and MPLS in myomectomy for the treatment of uterine fibroids.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with uterine fibroids before surgery on the basis of radiological or other examinations
* will consider TU-LESS or MPLS for myomectomy

Exclusion Criteria:

* patients reluctant to long-term follow-up

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Uterine fibroids occur only to female population
Enrollment: 5000 (Estimated)
Dates: Start 2023-06-24 (Actual); Primary Completion 2026-08-24 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Duration of hospital stay after surgery | From enrollment to 1 month after receiving myomectomy
  The number of days between myomectomy and the day of hospital discharge.

SECONDARY OUTCOMES:
VAS score at 4, 8, 12, 16, 20, 24 hours after myomectomy | From enrollment to 24 hours after myomectomy
  The visual analogue score at 4, 8, 12, 16, 20, 24 hours after myomectomy will be collected through questionnaire.
Time between myomectomy and exhaustion | From enrollment to 1 week after myomectomy.
  The exact time between myomectomy and exhaustion will be collected during wards round by directly asking the patients.
Time of surgery | From enrollment to 1 day after myomectomy.
  The time of surgery (from superficial incision to the end of umbilical suturing in experimental group and end of incision suturing in control group) will be collected during surgery.
Volume of bleeding during myomectomy | From enrollment to 1 day after myomectomy.
  The exact volume of bleeding during myomectomy in both experimental and control group will be collected during surgery.
Number of uterine fibroids resected during surgery. | From enrollment to 1 day after myomectomy.
  The exact number of uterine fibroids resected during myomectomy in both experimental and control group will be collected during surgery.
Pregnancy outcome | From enrollment to 2 years after myomectomy
  Whether the patient had pregnancy within 2 years after myomectomy. The information will be collected through online questionnaire and telephone.
Occurrence of pelvic and abdominal metastasis after myomectomy in cases with accidental uterine malignancy | From enrollment to 2 years after receiving myomectomy
  According to epidemiology data, a fraction of patients with primarily identified uterine fibroids will be pathologically diagnosed with uterine malignancy like uterine sarcoma after surgery. Whether the patients who were finally diagnosed with uterine malignancy based pathology developed abdominal or pelvic metastasis will be collected by telephone follow-up.

OTHER OUTCOMES:
Objective evaluation of incision healing | From enrollment to 3 months after myomectomy.
  The patients will be asked to give rating of the recovery of surgical incision from 1 (the most unsatisfied) to 10 (the most satisfied) through questionnaire and telephone follow up.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Second University Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided
We will share the study protocol after its publication

REFERENCES:
- [Result] Wright JD, Tergas AI, Burke WM, Cui RR, Ananth CV, Chen L, Hershman DL. Uterine pathology in women undergoing minimally invasive hysterectomy using morcellation. JAMA. 2014 Sep 24;312(12):1253-5. doi: 10.1001/jama.2014.9005. No abstract available. PMID 25051495
- [Result] Yuan P, Shan L, Yang X, Yu F, Ge Z, Wang M, Tan H. The merging of dual umbilical port-incisions for contained morcellation in laparoscopic myomectomy. Am J Obstet Gynecol. 2023 Jul;229(1):72-74. doi: 10.1016/j.ajog.2023.03.018. Epub 2023 Mar 17. PMID 36933684
- [Result] Glaser LM, Friedman J, Tsai S, Chaudhari A, Milad M. Laparoscopic myomectomy and morcellation: A review of techniques, outcomes, and practice guidelines. Best Pract Res Clin Obstet Gynaecol. 2018 Jan;46:99-112. doi: 10.1016/j.bpobgyn.2017.09.012. Epub 2017 Sep 29. PMID 29078975
- [Result] Wang L, Deng JY, Li KP, Zhu PY. A systematic review and meta-analysis comparing robotic single-site versus multi-port myomectomy. J Robot Surg. 2023 Aug;17(4):1319-1328. doi: 10.1007/s11701-023-01597-9. Epub 2023 Apr 24. PMID 37093509